CLINICAL TRIAL: NCT02611219
Title: Effect of Increased Activity on Deconditioning in Pediatric Stem Cell Transplant Recipients: A Feasibility Study
Brief Title: Deconditioning in Transplant
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201406031
Record Dates: First submitted 2015-11-12; First posted 2015-11-20 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Hematopoietic and Stem Cell Transplant
MeSH Terms: interventions — 2-methylcyclopentadienyl manganese tricarbonyl; Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Pediatric patients (Experimental): * Patients will wear a Fitbit Flex during hospitalization
  * Completion of Demographic Data Form at baseline, discharge from hospital, and at the six week clinic visit
  * Assist in recording time out of bed using the SCT Daily Activity Log
  * Fill out (some with help of parents) applicable questionnaires: Child Health Ratings Inventories-General Health Module (5-12 years), General Health Module-Baseline Adolescent-Self Report (13-18 years), General Health Module-Follow Up Adolescent-Self Report (13-18 years) at baseline, discharge from hospital, and at six week clinic visit
  * Patients will be assessed using standard physical therapy assessment tools to determine functioning, muscle strength, endurance, and mobility: The Functional Independence Measure for Children and Manual Muscle Testing is done weekly, discharge from hospital, and at six week clinic visit. The 3-Minute Step Test is done at admission, discharge from hospital, and at six week clinic visit.
  Interventions: Other: General Health Module-Baseline Adolescent-Self Report (13-18 years); Other: General Health Module-Follow Up Adolescent-Self Report (13-18 years); Other: Demographic Data Form; Other: SCT Daily Activity Log; Other: The Functional Independence Measure for Children; Other: Manual Muscle Testing; Other: 3-Minute Step Test; Other: HSCT Module-Follow Up Adolescent-Self Report (13-18 years); Other: HSCT Module-Follow Child-Self Report (5-12 years)
- Arm 2: Parents of pediatric patients (Experimental): * Parents will be considered participants as they will be completing study questionnaires.
  * Completion of Demographic Data Form at baseline
  * Assist in recording time out of bed using the SCT Daily Activity Log
  * Fill out applicable questionnaires: General Health Module-Baseline Parent Report -Adolescent (13-18 Years), General Health Module-Follow Up Parent Report-Adolescent (13-18 years), General Health Module-Baseline Parent Report-School Age (5-12 years), and General Health Module Follow Up Parent Report-School Age (5-12 years), HSCT Module-Follow UP Parent Report School Age (5-12 years), HSCT Module-Follow Up Parent Report Adolescent (13-18 years), HSCT Module-Follow Up Adolescent-Self Report (13-18 years), HSCT Module-Follow Child-Self Report (5-12 years) at baseline, discharge from hospital, and at six week clinic visit.
  * Assist child with Child Health Ratings Inventories-General Health Module (5-12 years) at baseline, discharge at hospital, and at six week clinic visit
  Interventions: Other: General Health Module-Baseline Parent Report-Adolescent (13-18 years); Other: General Health Module-Follow Up Parent Report-Adolescent (13-18 years); Other: General Health Module-Baseline Parent Report-School Age (5-12 years); Other: General Health Module-Follow Up Parent Report-School Age (5-12 years); Other: Demographic Data Form; Other: SCT Daily Activity Log; Other: HSCT Module-Follow Up Parent Report-adolescent (13-18 years); Other: HSCT Module-Follow Up Parent Report-School Age (5-12 years)

INTERVENTIONS:
Other: General Health Module-Baseline Adolescent-Self Report (13-18 years) — * 38 question questionnaire
  * Answers range from 1=all of the time to 5=none of the time
  Arms: Arm 1: Pediatric patients
Other: General Health Module-Follow Up Adolescent-Self Report (13-18 years) — * 38 question questionnaire about child
  * Answers range from 1=all of the time to 5=none of the time
  Arms: Arm 1: Pediatric patients
Other: General Health Module-Baseline Parent Report-Adolescent (13-18 years) — * 38 question questionnaire about child
  * 49 question questionnaire about parent
  * Answers range from 1-all of the time to 5=none of the time
  Arms: Arm 2: Parents of pediatric patients
Other: General Health Module-Follow Up Parent Report-Adolescent (13-18 years) — * 38 question questionnaire about child
  * 49 question questionnaire about parent
  * Answers range from 1-all of the time to 5=none of the time
  Arms: Arm 2: Parents of pediatric patients
Other: General Health Module-Baseline Parent Report-School Age (5-12 years) — * 34 question questionnaire about child
  * 49 question questionnaire about parent
  * Answers range from 1-all of the time to 5=none of the time
  Arms: Arm 2: Parents of pediatric patients
Other: General Health Module-Follow Up Parent Report-School Age (5-12 years) — * 34 question questionnaire about child
  * 49 question questionnaire about parent
  * Answers range from 1-all of the time to 5=none of the time
  Arms: Arm 2: Parents of pediatric patients
Other: Demographic Data Form — -16 questions about demographics such as household income, race, and gender
Other: SCT Daily Activity Log — * Uses Fitbit Flex
  * Log that lists time in 15 minute increments and allows for checking when out of bed and describing the activity that occurred while out of bed
Other: The Functional Independence Measure for Children — * 18-item, 7-level ordinal scale instrument that measures a child's consistent performance in essential daily functional skills. Three main domains (selfcare, mobility, and cognition) are assessed by interviewing or by observing a child's performance of a task to criterion standards
  * Categorized into 2 main functional streams: "Dependent" (ie, requires helper: scores 1-5) and "Independent" (ie, requires no helper: scores 6-7). Scores 1 (total assistance) and 2 (maximal assistance) belongs to the "Complete Dependence" category. Scores 3 (moderate assistance), 4 (minimal contact assistance), and 5 (supervision or set-up) belongs to the "Modified Dependence" category. Scores 6 (modified independence) and 7 (complete independence) belongs to the "Independent" category.
  Other Names: WeeFIM
  Arms: Arm 1: Pediatric patients
Other: Manual Muscle Testing — -Isometric muscle strength is tested in specific positions, usually with the muscle at an optimal working length. Using a "break" test, the test giver overpowers the muscle being tested to determine the muscle grade.
  Other Names: MMT
  Arms: Arm 1: Pediatric patients
Other: 3-Minute Step Test — * Using an aerobic step, the participant walks up and down for a given amount of time with the heart rate being checked before and after
  * Using the difference in heart rate and a shortness of breath scale, this test is able to give an estimate of aerobic tolerance
  Arms: Arm 1: Pediatric patients
Other: HSCT Module-Follow Up Adolescent-Self Report (13-18 years) — * 7 question questionnaire about child
  * Answers range from 1=all of the time to 5=none of the time
  Arms: Arm 1: Pediatric patients
Other: HSCT Module-Follow Child-Self Report (5-12 years) — * 10 question questionnaire about child
  * Answers range from 1=all of the time to 5=none of the time
  Arms: Arm 1: Pediatric patients
Other: HSCT Module-Follow Up Parent Report-adolescent (13-18 years) — * 7 question questionnaire about child
  * 49 question questionnaire about parent
  * Answers range from 1=all of the time to 5=none of the time
  Arms: Arm 2: Parents of pediatric patients
Other: HSCT Module-Follow Up Parent Report-School Age (5-12 years) — * 7 question questionnaire about child
  * 49 question questionnaire about parent
  * Answers range from 1=all of the time to 5=none of the time
  Arms: Arm 2: Parents of pediatric patients

SUMMARY:
The purpose of this feasibility study is to test the potential for successful implementation of an intervention designed to study the effect of six hours out of bed time on the overall level of deconditioning in pediatric stem cell transplant (SCT) patients. Previous research has demonstrated that deconditioning occurs rapidly over the course of the hospitalization post-transplant and can negatively impact quality of life. By encouraging patients to be out of bed for six hours each day, it is anticipated that patients will experience less deconditioning than those patients who previously had no established minimum time out of the bed.

ELIGIBILITY:
Inclusion Criteria (Pediatric Patients)

* Ages 7-17 years
* Admitted to hospital for stem cell transplant
* Speaks English

Inclusion Criteria (Parents of pediatric patients)

* Parents of children ages 7-17 years
* Parents of children admitted to hospital for stem cell transplant
* Speaks English

Exclusion Criteria (Pediatric Patients) -Admitted to transplant unit for autologous stem cell transplant, donor lymphocyte infusions, mesenchymal cell infusions, a second stem cell transplant, graft versus host disease or other complications post stem cell transplant will not be included

Exclusion Criteria (Parents of pediatric patients)

-Parents of children admitted to transplant unit for autologous stem cell transplant, donor lymphocyte infusions, mesenchymal cell infusions, a second stem cell transplant, graft versus host disease or other complications post stem cell transplant will not be included

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention of participants throughout the study | Baseline through 6 week clinic visit (up to an estimated 82 days)
  -Analyze the number of participants enrolled who continue through the 6 week clinic visit
Number of participants who achieve 6 hours out of bed through the 6 week clinic visit | Baseline through 6 week clinic visit (up to an estimated 82 days)
Quality of life as measured by General Health Module questionnaires | Discharge from hospital (estimated to be 40 days)
Quality of life as measured by General Health Module questionnaires | Baseline through 6 week clinic visit (up to an estimated 82 days)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Taylor, RN, BSN, CPHON, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu